CLINICAL TRIAL: NCT03221621
Title: Cost-effectiveness of Adalimumab With Adjuvant Surgery Versus Adalimumab Monotherapy in the Treatment of Hidradenitis Suppurativa'
Brief Title: Cost-effectiveness of Adalimumab and Surgery vs Adalimumab in HS
Acronym: HS-COST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Prothya Biosolutions (Industry)
Responsible Party: Principal Investigator, M.B.A. van Doorn, Principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-COST
Record Dates: First submitted 2017-07-04; First posted 2017-07-18 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: Acne inversa; Adalimumab; Cost-effectiveness
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: Patients will be treated with either the combination of adalimumab and surgery or adalimumab monotherapy for two years, both according to normal clinical practice. Patients on adalimumab monotherapy will be given the possibility to crossover into Group B when they do not achieve the HiSCR after 6 months of treatment. Additionally patients will be offered treatment with infliximab, according to clinical practice, until he last surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adalimumab Monotherapy (Active Comparator): Adalimumab injections will be administered through subcutaneously in a weekly dose of 40mg from week 4 up to 24 months (V8), after an initial dose of 160mg at week 0 and a 80mg dose at week 2, continued for 2 years in total.
  Interventions: Drug: Adalimumab Injection
- Adalimumab + Surgery (Experimental): Patients will be treated with a combination of adalimumab and wide excision, with a maximum of three surgical interventions within the first year. Adalimumab will be administered through subcutaneous injections in weekly dose of 40mg from week 4 up to 24 months (V8), after an initial dose of 160mg at week 0 and a 80mg dose at week 2, continued until the last surgery.
  Interventions: Procedure: Wide Excision; Drug: Adalimumab Injection

INTERVENTIONS:
Procedure: Wide Excision — Wide excision is performed under general anaesthesia or procedural sedation and analgesia (PSA). All lesional tissue, including fibrosis, is electrosurgically removed until the area is clear. The subcutaneous fat and epithelised sinus floors are left intact where possible. The wounds are left open to heal by secondary intention.
  Arms: Adalimumab + Surgery
Drug: Adalimumab Injection — Adalimumab will be administered through subcutaneous injections in weekly dose of 40mg from week 4 up to 24 months (V8), after an initial dose of 160mg at week 0 and a 80mg dose at week 2 until end of study or last surgery.
  Other Names: Humira

SUMMARY:
The primary objective of this randomized controlled clinical trial in a real life setting is to evaluate the cost-utility of limumab monotherapy compared with the combination of adalimumab and a maximum of three surgeries after two years of treatment in adult patients with moderate to severe HS.

DETAILED DESCRIPTION:
The primary objective of this randomized controlled clinical trial in a real life setting is to evaluate the cost-utility of limumab monotherapy (Group A) with the combination of adalimumab and a maximum of three surgeries (Group B) years of treatment in adult patients with moderate to severe HS.

Patients in group A will be treated with adalimumab monotherapy according to normal clinical practice and will be given the possibility to crossover into Group B when they do not achieve the HiSCR after 6 months of treatment. Additionally patients will be offered treatment with infliximab, according to clinical practice, until the last surgery. Patients in group B will receive adalimumab combined with a maximum of three adjuvant excisions of active lesions, both according to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Moderate to (very) severe HS defined as a score of ≥3 points on the PGA (range 1-5) and with a DLQI of at least 11 (range 0-30).
* Indication for adalimumab: i.e. uncontrolled disease (HS) under conventional therapy and/or minor surgery.
* A diagnosis of HS for more than six months prior to baseline.
* Clearance of HS can reasonably be achieved with three surgical interventions as based on consensus between two dermatosurgeons.
* Willing and able to undergo general anaesthesia or procedural sedation and analgesia.
* Able and willing to give written informed consent and to comply with the study requirements.

Exclusion Criteria:

* Contraindication for treatment with adalimumab (sepsis or risk of sepsis, active or latent tuberculosis, serious active local and/or chronic infections, heart failure NYHA class III/IV, severe liver disease, pre-existing HIV, active viral hepatitis, demyelinating disease, or allergy to adalimumab or any other ingredients of HUMIRA®).
* Previous or current use of adalimumab or other anti-TNF-α therapy.
* Current or recurrent clinically significant skin condition in the HS treatment area other than HS.
* Presence of other uncontrolled clinically significant major disease.
* Pregnant and lactating women.
* Malignancy (except basal cell carcinoma), lymphoproliferative disease or a history of malignancy.
* Current use of oral antibiotics (a washout period of 14 days is required).
* Current use of oral corticosteroids (a washout period of 30 days is required).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Cost-utility | 2 years
  Cost-utility: costs / point change in QALY

SECONDARY OUTCOMES:
Clinical efficacy using HiSCR | 2 years
  Assessment of clinical efficacy using HiSCR
Clinical efficacy using change in HS-PGA | 2 years
  Assessment of clinical efficacy using change in HS-PGA
Clinical efficacy using the number of flares | 2 years
  Assessment of clinical efficacy using the overall number of flares
Incidence and severity of treatment related adverse events | 2 years
  Assessment of tolerability and safety by recording the incidence and severity of all treatment related adverse events.
Cost-effectiveness | 2 years
  Cost-effectiveness: costs / point change in DLQI.
Quality of life using change in EQ-5D-5L | 2 years
  Assessment of changes in quality of life using the EuroQol-5D-5L (EQ-5D-5L)
Quality of life using change in DLQI | 2 years
  Assessment of changes in quality of life using the DLQI.
Quality of life using change in Skindex-17 | 2 years
  Assessment of changes in quality of life using the Skindex-17
Treatment satisfaction | 2 years
  Assessment of treatment satisfaction on a 5 point Likert scale
High sensitivity CRP | 2 years
  Assessment of change in high sensitivity CRP.
Cytokines | 3 months
  Assessment of cytokines as possible predictive biomarkers in skin biopsies.
Change in parameters of metabolic syndrome | 2 years
  Assessment of the change in parameters of metabolic syndrome: waist circumference, blood pressure, fasting plasma glucose, triglycerides, and HDL levels.
Change in parameters of pre-diabetes | 2 years
  Assessment of the change in parameters of pre-diabetes using a HOMA model
Identification of blood metabolite profiles | 3 months
  Identification of metabolites or metabolite profiles related to HS phenotypes, disease severity.
Identification of metabolites associated with treatment response | 3 months
  Identification of metabolites (or metabolite profiles) predicting clinical response to treatment.
Assessment of changes in metabolite (profiles) | 3 months
  Assessment of changes in metabolites (or metabolite profiles) in response to treatment.
Relation between adalimumab trough concentrations and treatment response | 3 months
  Relation between adalimumab trough concentrations and treatment response
Relation between adalimumab trough concentrations in serum and skin samples | 3 months
  Relation between adalimumab trough concentrations in serum and adalimumab trough concentrations in skin biopsies.
Influence of patient characteristics on adalimumab serum trough concentrations | 3 months
  adalimumab trough concentrations
Predictive value of early dry-blood-spots | 3 months
  Predictive value of early adalimumab concentrations using dry-blood-spots on treatment response at 3 months
Objectively assessed therapy adherence using adalimumab trough concentrations | 2 years
  Objectively assessed therapy adherence using adalimumab trough concentrations
Objectively assessed therapy adherence using collected syringes | 2 years
  Objectively assessed therapy adherence using collected syringes
Patient reported therapy adherence using a diary | 2 years
  Patient reported therapy adherence using a diary recording date of every injection.
Impact of surgery on quality of life measured with DLQI | 8 weeks after each surgery
  Assessment of the impact of wide excision on quality of life measured with DLQI
Impact of surgery on work productivity measured with WPAI | 8 weeks after each surgery
  Assessment of the impact of wide excision on work productivity and activity, measured with WPAI.
Wound closure time | through study completion, an average of 15 months
  Assessment of time to complete healing after wide excision using patient reported closure time.
Recurrence rate | through study completion, an average of 15 months
  Assessment of the recurrence of HS lesions after wide excision

CONTACTS AND LOCATIONS:
Overall Officials: Martijn van Doorn, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No